CLINICAL TRIAL: NCT01672450
Title: A Phase I Study of Intratumoral Injection of Interleukin-2 and Ipilimumab in Patients With Unresectable Stages III-IV Melanoma
Brief Title: A Study of Intratumoral Injection of Interleukin-2 and Ipilimumab in Patients With Unresectable Stages III-IV Melanoma
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: University of Utah (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: HCI56809
Record Dates: First submitted 2012-08-21; First posted 2012-08-24 (Estimated); Last update posted 2015-07-08 (Estimated); Status verified 2015-07

CONDITIONS: Melanoma
Keywords: Histologically or cytologically proven melanoma; Stages III-IV; accessible cutaneous, subcutaneous, and/or nodal lesions; ECOG performance status 0 to 2
MeSH Terms: conditions — Melanoma | interventions — Interleukin-2

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- All patients (Experimental): All participants in this study will receive the same treatment.
  Interventions: Drug: Intratumoral Ipilimumab and Interleukin-2

INTERVENTIONS:
Drug: Intratumoral Ipilimumab and Interleukin-2 — Only 1 lesion, 0.5 -2 cm, will be treated. Interleukin-2, 3 mIU IT TIW x 2 weeks (days 1, 3 and 5), then BIW x 6 weeks (days 1 and 4). Escalating doses of Ipilimumab (0.1, 0.25, 0.5, 1, 2, mg) IT weekly x 8 weeks

SUMMARY:
This is a single center, open phase I dose escalation study. This study will assess the highest tolerable intratumoral dose of ipilimumab (Yervoy) in combination with IL-2 (Proleukin) in patients with unresectable stages III-IV melanoma with accessible cutaneous, subcutaneous, and/or nodal lesions. The objective is to primarily assess the safety of the drug combination, and to secondarily obtain preliminary data on the clinical efficacy of the combination.

ELIGIBILITY:
Inclusion Criteria:

- Histological diagnosis of melanoma, unresectable stages III-IV with accessible cutaneous, subcutaneous, and/or nodal lesions , according to the AJCC Staging Manual, 7th Edition, 2011.

Note: Patients who are considered to have resectable disease but decline resection are eligible.

* At least one lesion > 0.5 cm and < 2 cm
* ECOG performance status 0, 1 or 2
* Negative pregnancy test for women of childbearing potential within 7 days of enrollment on study.
* WBC > 2,000/mm3; ANC > 1,000/mm3; platelet > 100,000/mm3;hemoglobin > 9 gm/dL (may be transfused)
* Serum bilirubin levels <1.5 mg/dL except for patients with Gilbert's syndrome.
* Serum aspartate transaminase (AST) and serum alanine transaminase (ALT) < 2.5 X upper limit of normal, alkaline phosphatase < 2.5 X upper limit of normal.
* Serum creatinine levels <1.5 mg/dL
* Women of childbearing potential should be advised to avoid becoming pregnant and men should be advised to not father a child while receiving treatment with ipilimumab or interleukin-2. Patients should agree to use an appropriate method of birth control while on study. Examples of adequate forms of birth control for women include oral or implanted contraceptives, intrauterine device (IUD), diaphragm with spermicide, cervical cap, abstinence, use of a condom by the sexual partner or sterile sexual partner and also based on the judgment of the investigator.
* Age > 18 years and of any gender or race.
* Able to provide informed consent and have signed an approved consent form that conforms to federal and institutional guidelines.

Exclusion Criteria:

* Concurrent therapy with any other non-protocol anti-cancer therapy
* Prior local therapy within 2 weeks or prior systemic therapy within 4 weeks of starting protocol treatment
* History of any other malignancy requiring active treatment
* Pre-existing autoimmunity: History of inflammatory bowel disease; history of symptomatic autoimmune disease (e.g., rheumatoid arthritis, systemic progressive sclerosis [scleroderma], systemic lupus erythematosus, autoimmune vasculitis [e.g., Wegener's Granulomatosis]); motor neuropathy considered of autoimmune origin (e.g., Guillain-Barre Syndrome). History of vitiligo is allowed.
* Chronic use immunosuppressants or systemic corticosteroids. Note: Chronic use is defined as requiring corticosteroids for greater than one month prior to enrollment on study. Corticosteroid use for less than 1 month prior to enrollment is allowed, but use must stop prior to starting study treatment.
* Clinically significant cardiovascular disease (e.g., uncontrolled hypertension [BP >150/100], myocardial infarction or stroke within 6 months, unstable angina), New York Heart Association (NYHA) Grade II or greater congestive heart failure, or serious cardiac arrhythmia requiring medication
* Currently active systemic infection
* Known history of HIV infection or chronic hepatitis B or C.
* The presence of any other medical or psychiatric disorder that, in the opinion of the treating physician, would contraindicate the use of the drugs in this protocol or place the subject at undue risk for treatment complications
* Pregnancy or breast feeding
* A history of a severe hypersensitivity reaction to ipilimumab or interleukin-2
* Any reason why, in the opinion of the investigator, the patient should not participate

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 12 (Actual)
Dates: Start 2012-09; Primary Completion 2014-08 (Actual); Study Completion 2014-08 (Actual)

PRIMARY OUTCOMES:
Number of Adverse Events per patient | 24 months
  To assess safety of interleukin-2 and Ipilimumab combination and to select the recommended dose regimen for future phase II studies

SECONDARY OUTCOMES:
Starting and Ending measurements of treated lesions | 24 months
  Clinical response rate of treated lesions
Starting and ending measurement of untreated lesions | 24 months
  Clinical response rate of untreated lesions

CONTACTS AND LOCATIONS:
Overall Officials: Hung Khong, MD, Principal Investigator — Huntsman Cancer Institute
Locations (1):
- Huntsman Cancer Institute, Salt Lake City, Utah, United States